CLINICAL TRIAL: NCT03608397
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multi-Center Trial to Evaluate the Efficacy and Safety of a Single Treatment of DaxibotulinumtoxinA for Injection in Adults With Isolated Cervical Dystonia (ASPEN-1)
Brief Title: Single Treatment of DaxibotulinumtoxinA for Injection in Adults With Isolated Cervical Dystonia (ASPEN-1)
Acronym: ASPEN-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Revance Therapeutics, Inc. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1720302
Record Dates: First submitted 2018-07-11; First posted 2018-08-01 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Cervical Dystonia
Keywords: DAXI; Cervical Dystonia; TWSTRS; Toxin
MeSH Terms: conditions — Torticollis | interventions — Botulinum Toxins, Type A; Injections

STUDY DESIGN:
Intervention Model Description: Approximately 300 subjects, recruited from study centers in the United States (US), Canada, and Europe will be randomized to DAXI high dose, DAXI low dose or placebo group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DAXI for injection low dose (Experimental): Low Dose Group
  Interventions: Biological: DaxibotulinumtoxinA for injection
- DAXI for injection high dose (Experimental): High Dose Group
  Interventions: Biological: DaxibotulinumtoxinA for injection
- Placebo (Placebo Comparator): Placebo Group
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: DaxibotulinumtoxinA for injection — DaxibotulinumtoxinA for injection is a sterile, white to off-white lyophilized product containing the active ingredient, daxibotulinumtoxinA, and inactive ingredients to be reconstituted with sterile, non-preserved, 0.9% sodium chloride solution saline.
  Arms: DAXI for injection high dose; DAXI for injection low dose
Biological: Placebo — Placebo is a sterile lyophilized product consisting of inactive ingredients without the neurotoxin to be reconstituted with sterile, non-preserved 0.9% sodium chloride solution.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel group, multi-center trial of two doses of daxibotulinumtoxinA (DAXI) for injection (high-dose; low-dose in adult subjects with isolated (primary) cervical dystonia (CD).

DETAILED DESCRIPTION:
Approximately 300 subjects, recruited from approximately 80 study centers in the United States (US), Canada, and Europe will be randomized to DAXI for injection high dose, DAXI for injection low dose, or placebo group, respectively. Subjects will be stratified by treatment center and history of prior treatment with botulinum neurotoxin (BoNT).

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18 to 80 years of age
* Meets diagnostic criteria for isolated CD (idiopathic; dystonic symptoms localized to the head, neck, shoulder areas) with at least moderate severity at Baseline (Day 1), defined as a TWSTRS-total score of at least 20, with at least 15 on the TWSTRS-Severity subscale, at least 3 on the TWSTRS-Disability subscale, and at least 1 on the TWSTRS-Pain subscale

Exclusion Criteria:

* Cervical dystonia attributable to an underlying etiology, (e.g., traumatic torticollis or tardive torticollis)
* Predominant retrocollis or anterocollis CD
* Significant dystonia in other body areas, or is currently being treated with BoNT for dystonia in areas other than those associated with isolated CD
* Severe dysphagia (Grade 3 or 4 on the Dysphagia Severity Scale) at Screening or Baseline (prior to study treatment)
* Any neuromuscular neurological conditions that may place the subject at increased risk of morbidity with exposure to BoNT, including peripheral motor neuropathic diseases (e.g., amyotrophic lateral sclerosis and motor neuropathy, and neuromuscular junctional disorders such as Lambert-Eaton syndrome and myasthenia gravis)
* Previous treatment with any BoNT product for any condition within the 14 weeks prior to Screening
* Botulinum Neurotoxin Type A (BoNTA), except the investigational daxibotulinumtoxinA, treatment-experienced subjects who had suboptimal or no treatment response to the most recent BoNTA injection for CD, as determined by the investigator, or history of primary or secondary non-response to BoNTA injections, known to have neutralizing antibodies to BoNTA; or have a history of botulinum toxin type B (rimabotulinumtoxinB [Myobloc/Neurobloc]) injection for CD due to non-response or suboptimal response to BoNTA

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2020-06-16 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS)-total score | Week 4 and Week 6
  TWSTRS is used to assess the severity of cervical Dystonia and the success of its treatment. The average of the change from baseline in TWSTRS-total score at Weeks 4 and 6 will be determined. TWSTRS-total score has a minimum score of 0 and a maximum score of 85, where higher scores represent worse outcomes. It is made up of the summation of 3 subscales: the Torticollis Severity Scale (minimum score of 0, maximum score of 35), the Disability Scale (minimum score of 0, maximum score of 30), and the Pain Scale (minimum score of 0, maximum score of 20).

SECONDARY OUTCOMES:
Change from Baseline TWSTRS-total score | Up to 36 Weeks
  Change from baseline in TWSTRS-total score (all post-treatment time points)
Duration of effect | Up to 36 Weeks
  Duration of effect based on target TWSTRS score
Patient Global Impression of Change (PGIC) Improvement | Week 4 or Week 6
  Percentage responders at Week 4 or 6
Incidence of treatment-emergent adverse events (Safety) | Up to 36 Weeks
  Evaluation of adverse events and serious adverse events over the course of the study.

OTHER OUTCOMES:
Change in TWSTRS subscale scores | Up to 36 Weeks
  Change from baseline in TWSTRS subscale scores (TWSTRS-Severity, TWSTRS-Disability, and TWSTRS-Pain) (all post-treatment time points)
Clinical Global Impression of Change (CGIC) | Up to 36 Weeks
  CGIC at all post-treatment time points
Patient Global Impression of Change (PGIC) | Up to 36 Weeks
  PGIC at all post-treatment time points

CONTACTS AND LOCATIONS:
Locations (75):
- United States (44):
  - HOPE Research Institute, Phoenix, Arizona
  - Movement Disorders Center of Arizona, Scottsdale, Arizona
  - The Parkinsons and Movement Disorder Institute, Fountain Valley, California
  - University of California, Irvine, Irvine, California
  - Loma Linda University, Loma Linda, California
  - USC Keck School of Medicine, Los Angeles, California
  - Care Access Research, Pasadena, California
  - Sutter Institute for Medical Research, Sacramento, California
  - Rocky Mountain Movement Disorders Center, Englewood, Colorado
  - Associated Neurologist, P.C., Danbury, Connecticut
  - New England Institute for Clinical Research, Stamford, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Design Neuroscience Center, Doral, Florida
  - University of Florida Center for Movement Disorders and Neurorestoration, Gainesville, Florida
  - Infinity Clinical Research, Hollywood, Florida
  - University of Florida Health Science Center Jacksonville, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Suncoast Neuroscience Associates, St. Petersburg, Florida
  - USF Parkinson's Disease and Movement Disorders Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Kansas Institute of Reseach, Overland Park, Kansas
  - Michigan State University, East Lansing, Michigan
  - QUEST Research Institute, Farmington, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - St Louis University, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Mount Sinai Movement Disorders Center, New York, New York
  - University of Rochester, Rochester, New York
  - Duke University, Durham, North Carolina
  - Wake Forest Health Sciences, Winston-Salem, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pennsylvania, Department of Neurology, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Coastal Neurology, Port Royal, South Carolina
  - Wesley Neurology Clinic, Cordova, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Neurology. P.A., Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Neurological Institute, Houston, Texas
  - Central Texas Neurology Consultants, Round Rock, Texas
  - University of Vermont Medical Center, Burlington, Vermont
- Austria (2):
  - Medical University Innsbruck, Innsbruck
  - Universitaetsklinik fuer Neurologie, Vienna
- University Health Network, Toronto Western Hospital, Toronto, Ontario, Canada
- Czechia (5):
  - Fakultni nemocnice Olomouc, Neurologicka klinika, Olomouc
  - Fakultní nemocnice Ostrava, Neurologicka klinika, Ostrava-Poruba
  - Lekarna Pardubicke nemocnice, Pardubice
  - Neurologicka klinika 1. LF UK a VFN v Praze, Prague
  - Vestra Clinics s.r.o., Rychnov nad Kněžnou
- France (4):
  - Hôpital Neurologique Pierre Wertheimer, Bron
  - CHU Grenoble Alpes, Grenoble
  - Hôpital Roger Salengro - CHRU de Lille, Lille
  - CHU Caremeau, Service de Neurologie, Nîmes
- Germany (6):
  - Praxis fuer Neurologie im Bismark Karrée, Berlin
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum rechts der Isar der TUM, München
  - GFO Kliniken Troisdorf, Betriebsstätte St. Johannes Sieglar, Troisdorf
  - Universitätsklinikum Tübingen, Tübingen
- Poland (6):
  - Szpital sw. Wojciecha Podmiot Leczniczy Copernicus Sp. Z o.o., Gdansk
  - Marta Dagmara BANACH Marta Banach Specjalistyczny Gabinet Neurologiczny, Krakow
  - Krakowska Akademia Neurologii, Krakow
  - Wojewodzki Szpital Specjalistyczny w Olsztynie, Olsztyn
  - Centrum Medyczne Pratia Warszawa, Warsaw
  - Mazowiecki Szpital Brodnowski Sp. z o.o., Warsaw
- Spain (4):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Burgos, Burgos
  - Hospital Universitario de La Princesa, Madrid
- United Kingdom (3):
  - Royal Devon and Exeter Foundation Trust Hospital, Exeter
  - The Walton Centre NHS Foundation Trust, Liverpool
  - Salford Royal NHS Foundation Trust, Salford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Comella CL, Jankovic J, Hauser RA, Patel AT, Banach MD, Ehler E, Vitarella D, Rubio RG, Gross TM; ASPEN-1 Study Group. Efficacy and Safety of DaxibotulinumtoxinA for Injection in Cervical Dystonia: ASPEN-1 Phase 3 Randomized Controlled Trial. Neurology. 2024 Feb 27;102(4):e208091. doi: 10.1212/WNL.0000000000208091. Epub 2024 Jan 31. PMID 38295339